CLINICAL TRIAL: NCT00431457
Title: Prospective Randomized Controlled Study of Neurostimulation in the Medial Temporal Lobe for Patients With Medically Refractory Medial Temporal Lobe Epilepsy; Controlled Randomized Stimulation Versus Resection (CoRaStiR)
Brief Title: Controlled Randomized Stimulation Versus Resection (CoRaStiR)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2007/005
Record Dates: First submitted 2007-02-02; First posted 2007-02-05 (Estimated); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Implantation intracranial electrode with immediate stimulation (Active Comparator)
  Interventions: Device: Implantation of an intracranial electrode
- Implantation intracranial electrode without stimulation (Placebo Comparator)
  Interventions: Device: Implantation of an intracranial electrode
- Resective surgery: amygddohyppocampertomy (Active Comparator)
  Interventions: Procedure: amygddohyppocampertomy

INTERVENTIONS:
Device: Implantation of an intracranial electrode — Implantation of an intracranial electrode will be followed.
  Arms: Implantation intracranial electrode with immediate stimulation; Implantation intracranial electrode without stimulation
Procedure: amygddohyppocampertomy — Resective surgery
  Arms: Resective surgery: amygddohyppocampertomy

SUMMARY:
Patients will be prospectively randomized to 3 different treatment arms:

* Treatment group 1: patients who undergo medial temporal lobe resection
* Treatment group 2: patients who receive immediate hippocampal neurostimulation
* Treatment group 3: patients who are implanted with an intracranial electrode but in whom hippocampal neurostimulation is delayed for 6 months.

Twelve months after inclusion unblinding will occur. Patients in group 2 and 3 will have the option to choose between continuing neurostimulation treatment or resective surgery.

Study visits will occur every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Presurgical candidates with pharmacoresistant partial seizures despite optimal medical treatment and history of temporal lobe epilepsy
* Age above 18 years
* TIQ > 80
* Able to give informed consent
* Average of 2 partial seizures per month during a baseline of 3 months. Recording of seizures must have been done in a prospective manner using standard seizure diaries.
* Able to adequately report seizure frequencies using standard seizure diaries
* Video-EEG characteristics showing temporal lobe seizure onset (left-sided or right-sided seizure onset) in at least one recorded habitual seizure
* Presence of a structural abnormality in the medial temporal lobe, suggestive of hippocampal sclerosis as evidenced by optimum MRI
* Women of child-bearing age will be required to use a reliable method of contraception during the study duration

Exclusion Criteria:

* Extratemporal epilepsy; multifocal epilepsy; evidence of bilateral medial temporal lobe epilepsy
* MR evidence of potentially epileptogenic lesions outside the medial temporal lobe such as dysplasias, tumours or cavernomas
* Prior resective intracranial surgery
* Patients who are candidates for invasive video-EEG recording or have previously been investigated with invasive video-EEG recording
* Patients who previously underwent any other type of neurostimulation for treating epilepsy
* Patients who are unable to fill in questionnaires and comply with protocol requirements
* Progressive neurological or medical conditions
* Medical or psychiatric conditions precluding surgery or compliance
* Patients taking antidepressant medication
* Pregnancy at study onset
* Previous (within the last 3 months), ongoing or planned participation in other treatment study protocols for epilepsy
* Contraindication for intracranial surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-06-01 (Actual); Primary Completion 2009-12-01 (Actual); Study Completion 2009-12-01 (Actual)

PRIMARY OUTCOMES:
To assess whether stimulation and/or resection produces a reduction in mean monthly seizure frequency that is greater than in the control group over 6 months of follow-up. | 6 months
To assess whether stimulation produces a reduction in mean monthly seizure frequency that is comparable to resection at 6 and 12 months of follow-up. | at 6 and 12 months of follow-up

SECONDARY OUTCOMES:
To assess whether stimulation yields better neuropsychological outcome compared to resection at 12 months of follow-up. | at 12 months of follow-up
responder rates during 3 month intervals | 3 months intervals
mean seizure free interval during 3 month intervals | 3 month intervals
seizure severity and seizure type during 3-month intervals | 3-month intervals
quality of life: changes in QOLIE 89 score at 6 and 12 months | at 6 and 12 months
mood assessment: changes in Beck depression scale scores at 6 and 12 month | at 6 and 12 month
Safety Objectives: | during twelve months after inclusion
Operative and postoperative complications and long-term side effects | during twelve months after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Paul Boon, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (3):
- University Hospital Ghent, Ghent, Belgium
- Germany (2):
  - UKB Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Freiburg, Freiburg im Breisgau

REFERENCES:
- [Derived] Chatzikonstantinou A. Epilepsy and the hippocampus. Front Neurol Neurosci. 2014;34:121-42. doi: 10.1159/000356435. Epub 2014 Apr 16. PMID 24777136
- See also: Website of the University Hospital Ghent — http://www.uzgent.be